CLINICAL TRIAL: NCT00349453
Title: Retrospective and Prospective Multicenter Study Using Deferiprone (L1) Alone or in Combination With Desferrioxamine for the Treatment of Iron Overload in Transfusion-dependent Patients
Brief Title: Study Using Deferiprone Alone or in Combination With Desferrioxamine in Iron Overloaded Transfusion-dependent Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lipomed (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DF-2/CH
Record Dates: First submitted 2006-07-06; First posted 2006-07-07 (Estimated); Last update posted 2011-12-12 (Estimated); Status verified 2011-12

CONDITIONS: Hemochromatosis
Keywords: Deferiprone; L1; Desferrioxamine; Hemochromatosis; Iron overload; Thalassemia
MeSH Terms: conditions — Hemochromatosis; Iron Overload; Thalassemia | interventions — Deferiprone; Long Interspersed Nucleotide Elements; Deferoxamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Deferiprone (L1) monotherapy (Experimental): Deferiprone (L1) monotherapy
  Interventions: Drug: Deferiprone (L1)
- Combination therapy (Experimental): Deferiprone (L1) and desferrioxamine combination treatment
  Interventions: Drug: Deferiprone (L1); Drug: Desferrioxamine

INTERVENTIONS:
Drug: Deferiprone (L1) — 50-100 mg/kg body weight daily
  Arms: Deferiprone (L1) monotherapy
Drug: Deferiprone (L1) — 75 mg/kg body weight daily
  Arms: Combination therapy
Drug: Desferrioxamine — 35-50 mg/kg body weight on 2 or more days per week
  Arms: Combination therapy

SUMMARY:
Systematical (retro- and prospective) investigation of the long-term safety (toxicity assessment according to CTCAE v3.0) and efficacy of deferiprone either given alone or in combination with desferrioxamine

DETAILED DESCRIPTION:
Patients with refractory anemias requiring regular blood transfusions accumulate iron at the rate of approximately 0.5 mg/kg/day, which may lead to serious organ toxicity, e.g. to the heart, liver and endocrine organs. The human body has no active mechanism for the excretion of excess iron. Therefore multiply transfused patients will develop a secondary hemosiderosis, if excess iron is not excreted by a chelating agent. Symptoms of iron-overload occur when body iron stores reach 10-20 g. At higher levels severe, even fatal complications, particularly cardiac failure, may develop.

Desferrioxamine (DFO, Desferal) is the established and commonly used iron-chelating drug, but is expensive and must be given by slow subcutaneous or intravenous infusion for 8-12 hours a day during 5-7 days weekly at a dosage of 40-50 mg/kg body weight/day. This often leads to failure of compliance of the patient and therefore to inefficient iron chelation. Further, some patients are hypersensitive to desferrioxamine and others suffer from toxicity, e.g. to the ears or eyes.

Deferiprone (L1; CP20; 1,2 dimethyl-3-hydroxypyrid-4-one) is an orally active iron chelator investigated in various clinical trials since 1987. Dosages of 75 - 100 mg/kg body weight/day of L1 have been considered effective to maintain stable iron balance (urinary iron excretion of 0.5 mg/kg/day) and to reduce serum ferritin levels between 6% and 25% within one year of treatment in iron-overloaded thalassemic patients. There exists long-term experience with patients who have received deferiprone continuously for more than 10 years so far. The main side effects encountered during a deferiprone therapy are arthropathy, gastrointestinal symptoms, headache, and mild zinc deficiency. These adverse reactions are usually reversed on reducing the dose or discontinuing the drug. Except for severe joint symptoms in few patients, most of the subjects in different clinical trials have been able to continue with L1 therapy for a long term. The most severe, but rare complication following administration of deferiprone is agranulocytosis or neutropenia.

A new treatment regimen combining deferiprone with desferrioxamine is currently being investigated in many countries. Preliminary data have demonstrated that the combined use of both drugs is highly active showing an additive or even synergistic effect (significant decrease of serum ferritin and hepatic iron content, increase of urinary iron excretion). This synergism could be explained by the different mode of action of the two drugs. It could be demonstrated that patients who were not sufficiently chelated with desferrioxamine or deferiprone, could achieve a negative iron balance with the combination treatment of both drugs. The combined regimen was generally well tolerated. It has been speculated that the individual toxicity profile of both drugs can be positively influenced by the simultaneous administration of L1 and DFO. The daily treatment with L1 tablets combined with at least twice a week administration of parenteral desferrioxamine is more patient-convenient and therefore may enhance the patient's compliance.

The primary aim of this study is to systematically investigate the long-term safety (toxicity assessment according to CTCAE v3.0) of deferiprone either given alone or in combination with desferrioxamine. Further, in patients agreeing to perform annual SQUID analysis of the liver, the annual change of liver iron concentration (LIC) will be examined for four years.

ELIGIBILITY:
Inclusion Criteria:

* Iron overloaded male or female patients with primary or secondary hemochromatosis
* Age: 4 years and older
* Patients with desferrioxamine toxicity or allergy (e.g. visual or hearing defects, bone abnormalities, reactions at injection site)
* Patients unable or unwilling to comply satisfactorily with regular desferrioxamine administration on 5-7 days/week
* Combination treatment: patients not sufficiently chelated with desferrioxamine or deferiprone monotherapy
* Patients must be willing to undergo routine screening including medical history, physical examination and hematology, biochemistry and other laboratory tests
* Written informed consent

Exclusion Criteria:

* Children under 4 years of age
* Female and male of reproductive age, sexually active but not taking adequate contraceptive precaution
* Woman who are pregnant or breast-feeding
* Patients with HIV
* Patients with active hepatitis requiring treatment
* Patients with severe hepatic failure, cirrhosis
* Patients with neutropenia (neutrophils less than 1.5 exp9/l, MDS: less than 0.5 exp9/l)
* Patients with thrombocytopenia (platelets less than 100 exp9/l, MDS: less than 20 exp9/l)
* Patients with decompensated heart failure (LVEF less than 40% or patients under continuous cardiac medication)
* Patients with severe renal failure

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2005-03; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Liver Iron Concentration (LIC) by SQUID | Yearly
Long-term safety profile | Long-term

SECONDARY OUTCOMES:
Serum ferritin | At quarterly control visits
Urinary Iron Excretion (UIE) | At six-monthly control visits
Heart iron content (optional) by MRI T2* and MRI SIR | Yearly

CONTACTS AND LOCATIONS:
Overall Officials: Petrign FG Töndury, MD, Principal Investigator; Markus Schmugge Liner, MD, Principal Investigator — University Children's Hospital, Zurich
Locations (13):
- Switzerland (13):
  - Cantonal Hospital, Children's Clinic, Aarau, Canton of Aargau
  - Cantonal Hospital, Aarau, Canton of Aargau
  - Private children's practice, Bern, Canton of Bern
  - Children's Hospital of Eastern Switzerland, Sankt Gallen, Canton of St. Gallen
  - University Children's Hospital, Zurich, Canton of Zurich
  - University Hospital, Zurich, Canton of Zurich
  - Private practice, Zürich (Kreis 11) / Oerlikon, Canton of Zurich
  - Private practice, Arzo, Canton Ticino
  - Private practice, Lugano, Canton Ticino
  - Regional Hospital, Lugano, Canton Ticino
  - Private practice, Riva San Vitale, Canton Ticino
  - Cantonal Hospital Graubünden, Chur, Kanton Graubünden
  - Private children's practice, Brig, Valais

REFERENCES:
- [Result] Tondury P, Zimmermann A, Nielsen P, Hirt A. Liver iron and fibrosis during long-term treatment with deferiprone in Swiss thalassaemic patients. Br J Haematol. 1998 Jun;101(3):413-5. doi: 10.1046/j.1365-2141.1998.00725.x. PMID 9633879
- [Result] Tondury P, Kontoghiorghes GJ, Ridolfi-Luthy A, Hirt A, Hoffbrand AV, Lottenbach AM, Sonderegger T, Wagner HP. L1 (1,2-dimethyl-3-hydroxypyrid-4-one) for oral iron chelation in patients with beta-thalassaemia major. Br J Haematol. 1990 Dec;76(4):550-3. doi: 10.1111/j.1365-2141.1990.tb07915.x. PMID 2265118